CLINICAL TRIAL: NCT05035849
Title: Comparison of the FGM Profiles in Patients of Type 2 Diabetes Treated With Sitagliptin and Acarbose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KY20190926-02
Record Dates: First submitted 2021-04-14; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Acarbose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients in group A were given sitagliptin and metformin for the first two weeks, and then were treated with acarbose and metformin for the second two weeks. FGM was used to monitor glycemic variations during the whole four weeks.
  Interventions: Drug: sitagliptin and acarbose
- Group B (Active Comparator): Patients in group B were given acarbose and metformin for the first two weeks, and then were treated with sitagliptin and metformin for the second two weeks.FGM was used to monitor glycemic variations during the whole four weeks.
  Interventions: Drug: sitagliptin and acarbose

INTERVENTIONS:
Drug: sitagliptin and acarbose — One group used first sitagliptin and metformin, then used acarbose and metformin. Another group used first acarbose and metformin, then used sitagliptin andmetformin.

SUMMARY:
The aim of the study is to compare the FGM glycemic profiles in patients with type 2 diabetes mellitus treated with sitagliptin and acarbose.

DETAILED DESCRIPTION:
In this study, 60 patients with type 2 diabetes were randomly divided into group A or group B after stable glucose control. Flash Glucose Mornitoring(FGM) will be used in patients with two groups. Patients in group A were given sitagliptin and metformin for the first two weeks, and then were treated with acarbose and metformin for the second two weeks. FGM was used to monitor glycemic variations during the whole four weeks. The opposite therapy was true for patients in group B.

ELIGIBILITY:
Inclusion Criteria:

1. Participate voluntarily and sign the subject informed consent before the test.
2. Patients with type 2 diabetes, aged 18-75 years, meeting the diagnostic criteria of WHO1999, have not been treated with any hypoglycemic drugs.
3. No acute complications such as diabetic ketoacidosis and diabetic hyperosmolar syndrome.
4. Subjects are able and willing to undergo FGM examination, diet and exercise regularly.

Exclusion Criteria:

1. Patients allergic to insulin.
2. Impaired liver and renal function, ALT 2.5 times higher than the upper limit of normal value;Serum creatinine was 1.3 times higher than the upper limit of normal.
3. A history of drug abuse and alcohol dependence within the past 5 years.
4. Systemic hormone therapy was used in recent 3 months.
5. Patients with poor compliance and irregular diet and exercise.
6. Patients with infection and stress within four weeks.
7. Patients who cannot tolerate flash glucose mornitoring(FGM).
8. Patients who are pregnant, nursing or preparing to become pregnant.
9. Any other apparent condition or comorption as determined by the investigator, such as severe heart and lung disease, endocrine disease, neurological disease, tumor disease, other pancreatic disease, history of mental illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Glycemic variations | Endpoint at the third month
  CV

SECONDARY OUTCOMES:
Glycemic variations | Endpoint at the third month
  TIR

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, MD, Study Chair — Nanjing First Hospital, Nanjing, Jiangsu, China, 210012
Locations (1):
- Gu Gao, Nanjing, China